CLINICAL TRIAL: NCT02763241
Title: Phase III Randomized Open-label Clinical Trial Comparing Cleanoze® Irrigation Device With Powder Preparation Versus Conventional Irrigation Method for Chronic Rhinitis
Brief Title: Cleanoze® Irrigation Device With Powder Preparation Versus Conventional Irrigation Method for Chronic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Farmaline Co.,Ltd., Thailand (Unknown)
Responsible Party: Principal Investigator, Patorn Piromchai, Assistance Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE581519
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis
Keywords: rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cleanoze® (Experimental): Cleanoze® consists of a powder made up of Sodium chloride and Sodium Bicarbonate. This powder when dissolved in 250 ml of water is closely resembles the content of a body fluid which normally baths the outside of the cells of the body. This fluid is isotonic solution.
  The patient will be instructed to use this isotonic solution for nasal irrigation daily.
  Interventions: Drug: Cleanoze®
- Syringe irrigation (Active Comparator): Nasal irrigation using sterile 0.9% NaCl 250 ml by 20 ml syringe
  The patient will be instructed to use this isotonic solution for nasal irrigation daily.
  Interventions: Drug: Saline (Syringe irrigation)

INTERVENTIONS:
Drug: Cleanoze® — Cleanoze® consists of a powder made up of Sodium chloride and Sodium Bicarbonate. This powder when dissolved in 250 ml of water is closely resembles the content of a body fluid which normally baths the outside of the cells of the body. This fluid is isotonic solution.
  Arms: Cleanoze®
Drug: Saline (Syringe irrigation) — Nasal irrigation using 250 ml normal saline pushing into the nostril by 20 ml syringe
  Arms: Syringe irrigation

SUMMARY:
The investigators proposed that the Cleanoze® is superior to the traditional nasal saline irrigation in term of the ease of use which will resulting in a better quality of life of the participants. This study will compared the efficacy, adverse reactions, complications and ease of use of Cleanoze® comparing with normal saline solution

DETAILED DESCRIPTION:
Cleanoze® consists of a powder made up of Sodium chloride and Sodium Bicarbonate. This powder when dissolved in 250 ml of water is closely resembles the content of a body fluid which normally baths the outside of the cells of the body. This fluid is isotonic solution.

The nasal saline irrigation is the common procedure for upper respiratory tract infection patients including chronic rhinitis. The physician usually order the normal saline with appropriate medication e.g. anti-histamines, nasal steroids and anti-biotics to treat this condition.

The investigators proposed that the Cleanoze® is superior to the traditional nasal saline irrigation in term of the ease of use which will resulting in a better quality of life of the participants. This study will compared the efficacy, adverse reactions, complications and ease of use of Cleanoze® comparing with normal saline solution.

Study Population: Any patients with chronic rhinitis (e.g. allergic rhinitis, vasomotor rhinitis) will be randomized to receive the study or control medication. The investigators will include the children 5 years and above which able to doing the lavage under the parents assistant or by them self.

Study Design: Phase III randomized controlled trial

Sample Size: Estimate from pilot study, the 71 patients per arm was estimated (142 participants totally).

Study Duration:

* Duration of enrollment is 1 year.
* The patients will be followed up to 1 months depend on the disease conditions.
* The data analysis will take 3 additional months
* The full report will complete after the data analysis within 3 months
* The total of 1 year and 6 months period needed for this study.

Primary Objective: To compare the satisfaction of the patients using Cleanoze® versus conventional device

Secondary Objective(s):

* The adherence to Cleanoze® device
* The durability of the Cleanoze® device
* The patient symptom score (VAS)
* The SNOT-22 questionaire for evaluating the quality of life of the patients

ELIGIBILITY:
Inclusion Criteria:

* Any patients with chronic rhinitis conditions regardless of any cause (e.g. allergic, irritant, infection)

Exclusion Criteria:

* Acute or chronic rhinosinusitis
* Acute nasopharyngitis (common cold)
* Patients with a tendency to aspirate such as cerebrovascular accident, cranio-facial diseases.
* Sinunasal, nasopharyngeal and skull base tumors
* Age under 5 years old.
* Cannot administer a saline irrigation under the assistant of a care giver.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction score | 1 month
  This score will be evaluated at the end of 1 month using using the satisfaction questionaire

SECONDARY OUTCOMES:
The adherence to Cleanoze® devic | 1 month
  The adherence will be evaluated by the diary that the investigator given to the participants
The durability of the Cleanoze® device | 1 month
  The durability will be evaluated by inspecting the device at the end of 1 month period
The symptoms score of the patients | 1 month
  The symptoms score will be evaluated using the one-question VAS scale
The Sino-Nasal Outcome Test-22 Questionnaire (SNOT-22) score | 1 month
  The SNOT-22 score will be evaluated by using SNOT-22 questionnaire
Adverse events | 1 month
  The adverse events will be recorded in the case record form at follow-up time

CONTACTS AND LOCATIONS:
Overall Officials: Patorn Piromchai, MD, MSc, Principal Investigator — Khon Kaen University
Locations (1):
- Department of Otolaryngology, Khonkaen University, Muang, Khonkaen, Thailand

IPD SHARING:
Plan to Share IPD: No